CLINICAL TRIAL: NCT01585467
Title: Selective Radiography in Anterior Shoulder Dislocation: Prospective Validation Rule of Decision Rules Derived in Fresno and Quebec
Brief Title: Anterior Shoulder Dislocation
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 02102010
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Shoulder Dislocation
Keywords: Anterior Shoulder Dislocation; Shoulder Dislocation; Shoulder Pain; Shoulder Deformity
MeSH Terms: conditions — Shoulder Dislocation; Shoulder Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To compare and validate the two clinical algorithms

DETAILED DESCRIPTION:
Clinical Decision rules have safely and successfully allowed clinicians to reduce the total number of radiographs ordered, while detecting patients with important pathology or injuries. The Ottawa Ankle and Knee Rules were developed from a series of studies, and have successfully reduced the number of radiographs ordered by physicians without missing serious ankle fractures (1-4). Likewise, the NEXUS group developed a clinical decision rule for the selection of blunt trauma patients who are appropriate for imaging, based on clinical features (5).

Drs. Hendey and Emond have separately developed similar algorithms for selective radiography in patients with a suspected shoulder dislocation (6-10). The goal of the current study is to compare and validate the two clinical algorithms.

Both approaches examine clinical features that are readily accessible to the physician at the time of ED evaluation. In the pre-reduction assessment, both algorithms included the mechanism of injury and whether the patient had experienced a previous shoulder dislocation. Hendey additionally assessed whether the physician was clinically confident of the dislocation (8). Emond additionally included the age of the patient, and the presence or absence of humeral ecchymosis (9). In the post-reduction assessment, both algorithms emphasize the importance of clinical certainty of reduction, as well as the presence of a fracture dislocation.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 18 years and older
* patient with a suspected acute anterior shoulder dislocation

Exclusion Criteria:

* patients under 18 years of age
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Prospective validation of clinical decision rules | to be measured at study conclusion

CONTACTS AND LOCATIONS:
Locations (2):
- University of California, San Francisco-Fresno, Fresno, California, United States
- Universite Laval Pavillon Ferdinand-Vandry, Qubec, Quebec, Canada

REFERENCES:
- [Background] Stiell IG, McKnight RD, Greenberg GH, McDowell I, Nair RC, Wells GA, Johns C, Worthington JR. Implementation of the Ottawa ankle rules. JAMA. 1994 Mar 16;271(11):827-32. PMID 8114236
- [Background] Stiell IG, Greenberg GH, McKnight RD, Nair RC, McDowell I, Reardon M, Stewart JP, Maloney J. Decision rules for the use of radiography in acute ankle injuries. Refinement and prospective validation. JAMA. 1993 Mar 3;269(9):1127-32. doi: 10.1001/jama.269.9.1127. PMID 8433468
- [Background] Stiell IG, Wells GA, Vandemheen KL, Clement CM, Lesiuk H, De Maio VJ, Laupacis A, Schull M, McKnight RD, Verbeek R, Brison R, Cass D, Dreyer J, Eisenhauer MA, Greenberg GH, MacPhail I, Morrison L, Reardon M, Worthington J. The Canadian C-spine rule for radiography in alert and stable trauma patients. JAMA. 2001 Oct 17;286(15):1841-8. doi: 10.1001/jama.286.15.1841. PMID 11597285
- [Background] Stiell IG, Greenberg GH, Wells GA, McDowell I, Cwinn AA, Smith NA, Cacciotti TF, Sivilotti ML. Prospective validation of a decision rule for the use of radiography in acute knee injuries. JAMA. 1996 Feb 28;275(8):611-5. PMID 8594242
- [Background] Hoffman JR, Mower WR, Wolfson AB, Todd KH, Zucker MI. Validity of a set of clinical criteria to rule out injury to the cervical spine in patients with blunt trauma. National Emergency X-Radiography Utilization Study Group. N Engl J Med. 2000 Jul 13;343(2):94-9. doi: 10.1056/NEJM200007133430203. PMID 10891516
- [Background] Hendey GW, Kinlaw K. Clinically significant abnormalities in postreduction radiographs after anterior shoulder dislocation. Ann Emerg Med. 1996 Oct;28(4):399-402. doi: 10.1016/s0196-0644(96)70004-5. PMID 8839524
- [Background] Hendey GW. Necessity of radiographs in the emergency department management of shoulder dislocations. Ann Emerg Med. 2000 Aug;36(2):108-113. doi: 10.1067/mem.2000.108314. PMID 10918101
- [Background] Hendey GW, Chally MK, Stewart VB. Selective radiography in 100 patients with suspected shoulder dislocation. J Emerg Med. 2006 Jul;31(1):23-8. doi: 10.1016/j.jemermed.2005.09.006. PMID 16798149
- [Background] Emond M, Le Sage N, Lavoie A, Moore L. Refinement of the Quebec decision rule for radiography in shoulder dislocation. CJEM. 2009 Jan;11(1):36-43. doi: 10.1017/s1481803500010903. PMID 19166638
- [Background] Emond M, Le Sage N, Lavoie A, Rochette L. Clinical factors predicting fractures associated with an anterior shoulder dislocation. Acad Emerg Med. 2004 Aug;11(8):853-8. doi: 10.1111/j.1553-2712.2004.tb00768.x. PMID 15289192